CLINICAL TRIAL: NCT05837702
Title: Comparison of the Effects of Erector Spina Plan Block and Paravertebral Block in Laparoscopic Cholecystectomies on Pain Management.
Brief Title: Pain Management in Laparoscopic Cholecystectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Elvan Yilmaz, Assistant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021/ 283
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Nerve Block
Keywords: Erector Spinae Plane Block; Paravertebral Block; Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector Spinae Plane Block (ESPB) (Experimental): The spinous processes of the vertebrae were marked up to T8 level. After providing antisepsis of the skin with 10% povidone iodine, the ultrasound probe was placed at T8 level parallel to the vertebral spine at T8. The transverse process (TP) and hyperechoic pleura were observed 2.5cm right lateral of the spinous process. Using the in-plane approach, the needle was placed in the caudal direction. After confirming displacement of the pleura with 0.5-1ml local anaesthetic (LA), 20ml 0.25% bupivacaine was administered for the block .
  Interventions: Procedure: ESPB
- Paravertebral Block (PVB) (Active Comparator): After sterilisation of the skin with povidone iodine, the probe covered with a sterile sheath was placed 3cm lateral of the T8 spinous process. The trapezius, rhomboid major, and erector spinae muscles, and the TP of the vertebrae were visualised. The needle was placed craniocaudally within the fascial plane of the deep surface of the erector spina muscle above the bone shadow of the TP. The fluid dissemination was confirmed by raising the placement of the needle tip towards the erector spina muscle. 20ml 0.25% bupivacaine was applied to this region and the spread of local anaesthetic was observed
  Interventions: Procedure: PVB
- Control (Active Comparator): No block has been done
  Interventions: Procedure: CONTROL

INTERVENTIONS:
Procedure: ESPB — Erector spinae plane block
  Arms: Erector Spinae Plane Block (ESPB)
Procedure: PVB — Paravertebral Block
  Arms: Paravertebral Block (PVB)
Procedure: CONTROL — No block has been done
  Arms: Control

SUMMARY:
Erector spinae plane (ESP) block is a more recent method than paravertebral block (PVB) and has a lower risk of complications. The aim of this study was to compare postoperative analgesia requirements and side-effects in terms of safely reaching the maximum analgesic effect in patients.

DETAILED DESCRIPTION:
The primary aim of this study was to compare ESP block and PVB as important postoperative pain management in terms of being able to reliably reach the highest analgesic efficacy in patients who underwent laparoscopic surgery which is a frequently applied surgery. The secondary aim was to determine the incidence of postoperative nausea, vomiting and side-effects, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* aged >18 years
* patients with the American Society of Anesthesiologists (ASA) physical status I/II -who were planned to undergo laparoscopic cholecystectomy surgery

Exclusion Criteria:

* Did not provide informed consent,
* Had any psychiatric or mental problem that prevented understanding of the informed consent form
* They were planned to undergo emergency cholecystectomy,
* Had any allergy or hypersensitivity to local anaesthetic,
* Had an infection in the needle entry area
* History of coagulopathy or the use of anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Total tramadol consumption | 24 hours postoperatively
  Consumption at the end of 24 hours will be monitored by planning a 10mg bolus, a 10-minute lock-in time, through a patient-controlled analgesia device.

SECONDARY OUTCOMES:
Visual analog scale (VAS) at rest and when coughing | at 0, 5, 10,20 minutes and 1, 2,4 , 6, 12 and 24 hours postoperatively
  11-point scale where 0=no pain and 10=worst pain
Analgesic drug consumption other than tramadol | 24 hours postoperatively
  in mg
Heart Rate | preoperative, after insufflation, after exsufflation, after extubation( 5,10,20,30 minutes)
  beats /min
Mean arterial pressure (MAP) | preoperative, after insufflation, after exsufflation, after extubation( 5,10,20,30 minutes)
  mm-hg
Incidence of postoperative nausea & vomiting (PONV) | 24 hours postoperatively
  Number of patients developing PONV
Shoulder pain | 24 hours postoperatively
  Number of patients developing shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: elvan tekir yilmaz, Study Director — Giresun University
Locations (1):
- Giresun University Medical School Hospital., Giresun, Merkez, Turkey (Türkiye)